CLINICAL TRIAL: NCT00670176
Title: Pre- and Postoperative Cardiopulmonary Rehabilitation Reduces Complications After Coronary Artery Bypass Surgery: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Sul de Santa Catarina (Other Government)
Collaborators: ICSC (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICSC01
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Bypass Surgery
MeSH Terms: interventions — Rehabilitation; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Behavioral: REHAB (Pre- and postoperative cardiopulmonary rehabilitation)

INTERVENTIONS:
Behavioral: REHAB (Pre- and postoperative cardiopulmonary rehabilitation)

SUMMARY:
Pre- and postoperative cardiopulmonary rehabilitation reduces complications after coronary artery bypass surgery. This study was conducted as a randomized trial to verify this hypothesis in our institution. ICSC

ELIGIBILITY:
Inclusion Criteria:

* All CAB patients

Exclusion Criteria:

* SCA in the previous 24h and incapacity of doing light exercise. Valvular patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56
Dates: Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
length of stay in the ICU (in minutes); days on the ward after ICU until hospital discharge; pneumonia with the need for antibiotic treatment; and atrial fibrillation or flutter detected on daily-performed electrocardiograms

SECONDARY OUTCOMES:
time until oro-tracheal tube (OTT) removal, occurrence of pleural effusion, atelectasis, change in peak-flow (baseline vs. 2 hours after extubation vs. discharge), and changes in the 6-minute-walking distance between enrollment and hospital discharge.